CLINICAL TRIAL: NCT06525480
Title: Pulmonary Thromboembolism in Patients Undergoing Percutaneous Pulmonary Thrombectomy: Need for Mechanical Respiratory And/or Circulatory Assistance
Brief Title: Mechanical Respiratory/circulatory Support in Patients with Pulmonary Thrombectomy
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)102/202
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Embolism and Thrombosis; Extracorporeal Membrane Oxygenation; Percutaneous Pulmonary Thrombectomy
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Percutaneous pulmonary thrombectomy — Pulmonary thrombus extraction

SUMMARY:
Pulmonary embolism (PE) results from embolization of venous thrombi in the branches of the pulmonary arteries.

Although anticoagulation is usually the preferred method of treatment, patients with high-risk and/or intermediate/high-risk pulmonary embolism may benefit from immediate reperfusion therapy, such as mechanical catheter thrombectomy. During this procedure, there may be an increase in pulmonary pressures caused by the introduction of pulmonary catheters, which may trigger hemodynamic instability. In addition, anesthesia performed during percutaneous mechanical thrombectomy may precipitate hemodynamic and respiratory compromise due to hypoxia, hypercapnia and increased airway pressure.

We will perform a retrospective, single-center study to determine the incidence and immediate causes of hemodynamic and/or respiratory deterioration, before, during and after (first 30 days) of percutaneous pulmonary thrombectomy, as well as the need for mechanical respiratory/circulatory support.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a consequence of the embolization of venous thrombi in the branches of the pulmonary arteries. It affects approximately 1 in 1,000 people per year worldwide and represents the third cause of cardiovascular death.

The degree of hemodynamic compromise due to PE can be determined by imaging studies, such as computed tomography angiography, transthoracic echocardiography (TTE), and transesophageal echocardiography (TEE). Additionally, laboratory tests may suggest circulatory compromise, such as elevated levels of cardiac troponin and N-terminal pro b-type natriuretic peptide (NT-proBNP) at the time of PE presentation.

There are different classifications to evaluate the severity of PE and we consider the presence of hemodynamic instability to differentiate high-risk PE from intermediate-risk PE. The presence of hemodynamic instability includes a state of obstructive shock (signs of hypoperfusion associated with a systolic blood pressure (SBP) <90mmHg, and/or SBP ≥ 90mmHg with the need for vasoactive drugs), persistent hypotension (SBP<90mmHg for ≥ 15 min or SBP decrease ≥ 40mmHg compared to baseline) or cardiac arrest with the need for cardiopulmonary resuscitation (CPR). The high risk of PE also includes the existence of some parameter included in the sPESI such as: history of cancer, age over 80 years, heart rate ≥ 110 bpm, history of chronic obstructive pulmonary disease, SBP <100 mmHg and SpO2 <90%.

Patients with high-risk and/or intermediate/high-risk pulmonary embolism benefit from immediate reperfusion therapy, such as systemic thrombolysis, catheter-directed thrombolysis, catheter thrombectomy or surgery. Although the incidence of complications and mortality in high-risk PE patients has been determined, the incidence and immediate causes of hemodynamic and/or respiratory deterioration before, during, and after pulmonary thrombectomy are unknown. Pulmonary thrombectomy is a technique that consists of the extraction or dissolution, using endovascular devices, of the thrombus that partially or totally obstructs a pulmonary artery. It is generally associated with the local intra-thrombus administration of thrombolytic drugs. The increase in pulmonary intravascular pressure generated during the procedure can trigger the appearance of complications (arrhythmias, acute overload of the right ventricle, hemodynamic and/or respiratory instability, shock, cardiovascular arrest). These complications usually require an increase in hemodynamic support (with an increase in vasoactive drugs) and/or respiratory support (orotracheal intubation and mechanical ventilation), and even mechanical support with ECMO, usually veno-arterial ECMO for cardiovascular assistance. Also, the type of anesthesia performed can precipitate the hemodynamic and/or respiratory compromise of patients due to the possible presence of hypoxia and hypercapnia in patients who present hypoventilation, and the increase in airway pressures caused by orotracheal intubation and mechanical ventilation. In some cases, the use of mechanical circulatory support, usually ECMO, may be justified; but it is currently unclear whether VA-ECMO should be initiated in all high-risk PE patients. It must be considered that VA-ECMO is associated with innumerable complications (bleeding, thrombi, vascular complications), which increase the longer the duration of support.

Determining the incidence and causes or context of the onset of hemodynamic and/or respiratory deterioration (leading to shock, need for orotracheal intubation, cardiopulmonary arrest and/or mechanical support with ECMO), before, during and after thrombectomy pulmonary disease, could help reduce the morbidity and mortality of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with high/intermediate risk of pulmonary embolism who undergo pulmonary mechanical thrombectomy

Exclusion Criteria:

* Patients under 18 years of age
* Low-risk pulmonary embolism patients
* Patients who do not undergo pulmonary mechanical thrombectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with intermediate/high risk pulmonary thromboembolism requiring percutaneous pulmonary thrombectomy
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence and causes of hemodynamic and/or respiratory instability | From the diagnosis of pulmonary embolism until 30 days after percutaneous pulmonary thrombectomy
  Determine the incidence and immediate causes of hemodynamic and/or respiratory instability in patients with intermediate/high risk of pulmonary embolism.
  * Hemodynamic instability: obstructive shock (signs of hypoperfusion associated with a systolic blood pressure (SBP) <90mmHg, and/or SBP ≥ 90mmHg with the need for vasoactive drugs), persistent hypotension (SBP<90mmHg for ≥ 15 min or SBP decrease ≥ 40mmHg compared to baseline) or cardiac arrest with the need for cardiopulmonary resuscitation
  * Respiratory instability: SpO2 <90%, dyspnea

SECONDARY OUTCOMES:
Need for ECMO treatment | From the diagnosis of pulmonary embolism until 30 days after percutaneous pulmonary thrombectomy
  Determine the percentage of patients who require ECMO and its associated complications (hemorrhage, thrombosis, ischemia)

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d´Hebron Research Institute VHIR, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No